CLINICAL TRIAL: NCT06326684
Title: Influence of Orexin Antagonism on Motivation for Alcohol
Brief Title: Suvorexant and Alcohol
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 88524; R01AA030775 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will be treated daily with an oral placebo.
  Interventions: Drug: Alcohol; Drug: Placebo
- Suvorexant Dose 1 (Experimental): Subjects will be treated daily with oral suvorexant (10 mg).
  Interventions: Drug: Alcohol; Drug: Suvorexant
- Suvorexant Dose 2 (Experimental): Subjects will be treated daily with oral suvorexant (20 mg).
  Interventions: Drug: Alcohol; Drug: Suvorexant

INTERVENTIONS:
Drug: Alcohol — The pharmacodynamic effects of alcohol (0.2 and 0.4 g/kg) will be determined.
Drug: Placebo — The effects of placebo will be determined.
  Arms: Placebo
Drug: Suvorexant — The effects of suvorexant dose 1 will be determined.
  Arms: Suvorexant Dose 1
Drug: Suvorexant — The effects of suvorexant dose 2 will be determined.
  Arms: Suvorexant Dose 2

SUMMARY:
This research will translate findings from preclinical research and provide the initial clinical evidence that orexin antagonism reduces motivation for alcohol, as well as other alcohol-associated maladaptive behaviors in people with Alcohol Use Disorder. This study will also provide basic science information about the orexinergic mechanisms underlying the pharmacodynamic effects of alcohol in humans. As such, the outcomes will contribute to our understanding of the clinical neurobiology of Alcohol Use Disorder. Overall, the proposed work seeks to expand the scope of current clinical neuroscience research on alcohol addiction by focusing on orexin, which has strong preclinical evidence supporting its critical role in addiction but remains unstudied in humans.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

1. Able to speak and read English.
2. Not seeking treatment at the time of the study.
3. Between the ages of 21 and 55 years.
4. Engaging in at least one binge drinking episode, per the NIAAA definition, in the last 30 days.
5. Fulfillment of moderate or severe DSM-5 diagnostic criteria for AUD based on computerized SCID results reviewed by a psychiatrist or psychologist.
6. ECG, read by cardiologist, within normal limits.
7. Body mass index of 19 - 35.
8. Birthing individuals using an effective form of birth control and not pregnant or breast feeding.
9. Judged by the medical staff to be psychiatrically and physically healthy (i.e., no current severe SUD or psychiatric diagnoses other than AUD or Tobacco Use Disorder; no current physical diagnoses that would interfere with study participation according to study physician judgment).
10. Not currently physiologically dependent on any substances.
11. Able to abstain from alcohol during admission (i.e., not physically dependent on alcohol and scores less than 8 on Clinical Institute Withdrawal Assessment for Alcohol [CIWA-Ar] at screening).
12. Not currently taking any prescribed medications for a chronic condition (other than birth control).
13. No indication of sleep apnea on the STOP-Bang questionnaire (score of 5 or greater).
14. No contraindications/allergies to suvorexant.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All gender identities are eligible.
Enrollment: 30 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Reinforcing Effects of Alcohol | 6 times over approximately 3 week inpatient admission.
  Number of Times Subjects Choose Alcohol (Maximum of 5 Choices) Over Money

SECONDARY OUTCOMES:
Craving | 6 times over approximately 3 week inpatient admission.
  Subjects will report their craving during 6 sessions while they are admitted to our inpatient unit. Measured using a 10 point craving questionnaire with higher scores meaning greater craving.
Mood | 6 times over approximately 3 week inpatient admission.
  Subjects will complete the Profile of Mood States during 6 sessions while they are admitted to our inpatient unit. Scores range from 0 to 4 with higher scores indicating stronger mood.
Alcohol Response | 6 times over approximately 3 week inpatient admission.
  Subjects will complete the Biphasic Alcohol Effects Scale during 6 sessions while they are admitted to our inpatient unit. Scores range from 0 to 10 with higher scores indicating greater responses.
Heart rate | Daily over approximately 3 week inpatient admission.
  Beats per minute. Measured daily during inpatient admission.
Blood pressure | Daily over approximately 3 week inpatient admission.
  mm Hg. Measured daily during inpatient admission.
Breath Alcohol Level | Daily over approximately 3 week inpatient admission.
  Percent. Measured daily during inpatient admission.
Temperature | Daily over approximately 3 week inpatient admission.
  Degrees Fahrenheit. Measured daily during inpatient admission.
Side Effects | Daily over approximately 3 week inpatient admission.
  Subjects will complete a side effects questionnaire daily while they reside on the inpatient unit. Side Effects questions will query subjects about common effects of centrally active medications.
Delay Discounting | 6 times over approximately 3 week inpatient admission.
  Subjects will complete the delay discounting task during 6 sessions while they are admitted to our inpatient unit. Responses will be used to calculate discounting slope (i.e., K).
n-back Task | 6 times over approximately 3 week inpatient admission.
  Subjects will complete the n-back task during 6 sessions while they are admitted to our inpatient unit. Percentage of correct responses will be the outcome.
Stop-Signal Task Inhibitory Failures | 6 times over approximately 3 week inpatient admission.
  Subjects will complete the stop-signal task during 6 sessions while they are admitted to our inpatient unit. Proportion of inhibitory failures will be the outcome variable.
Sleep | Daily over approximately 3 week inpatient admission.
  Subjects will complete the St. Mary's Sleep Questionnaire daily while they are admitted to our inpatient unit. Total sleep time will be the outcome variable and will be recorded in minutes. Higher scores indicate more sleep. Total sleep time is measured by self-report; minimum score=0, maximum score=1440 per day.

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Psychopharmacology of Addiction Laboratory, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No